CLINICAL TRIAL: NCT06213519
Title: The Efficacy and Safety of Hyperthermic Intraperitoneal Chemotherapy （HIPEC）Combined With SOX and Sintilimab in the Treatment of Advanced Gastric Cancer With Peritoneal Metastasis: A Prospective, Single-arm, Phase II Clinical Study
Brief Title: HIPEC Combined With SOX and Sintilimab in the Treatment of Advanced Gastric Cancer With Peritoneal Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Bo Zhang, MD, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH-2023-1784
Record Dates: First submitted 2024-01-01; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Peritoneal Metastases; Gastric Cancer
Keywords: gastric cancer; peritoneal metastasis; HIPEC; first-line
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX+sintilimab+HIPEC (Experimental): Patient will receive SOX regimen (oxaliplatin 100mg/m2, d1, S-1 BSA<1.25m2 40mg, twice a day; 1.25m2 ≤ BSA < 1.5m2 50mg, twice a day; BSA ≥ 1.5m2 60mg, twice a day; d1-14) chemotherapy combined with sintilimab (200mg, d1), once every three weeks. In the first cycle, HIPEC (paclitaxel 80 mg/m2, d1-d3) will be administrated, and HIPEC or intraperitoneal chemotherapy (paclitaxel 80 mg/m2, d1) will be administrated in the second and third cycles according to the patient's condition. Then, another 3-cycle SOX regimen of systemic chemotherapy. After the end of 6 cycles, maintain treatment with a combination of S-1 and sintilimab until disease progression or intolerable toxicity.
  Interventions: Drug: S-1, Oxaliplatin sintilimab HIPEC

INTERVENTIONS:
Drug: S-1, Oxaliplatin sintilimab HIPEC — 1. Exploratory laparoscopy or laparotomy
  2. SOX regimen (oxaliplatin 100mg/m2, d1, S-1 BSA<1.25m2 40mg, twice a day; 1.25m2 ≤ BSA < 1.5m2 50mg, twice a day; BSA ≥ 1.5m2 60mg, twice a day; d1-14) chemotherapy combined with sintilimab (200mg, d1), once every three weeks.
  3. In the first cycle, HIPEC (paclitaxel 80 mg/m2, d1-d3) will be administrated,
  4. In the second and third cycles, HIPEC or intraperitoneal chemotherapy (paclitaxel 80 mg/m2, d1) will be administrated according to the patient's condition.
  5. Another 3-cycle SOX regimen of systemic chemotherapy.
  6. After the end of 6 cycles, maintain treatment with a combination of S-1 and sintilimab until disease progression or intolerable toxicity.

SUMMARY:
The prognosis of patients with peritoneal metastasis from gastric cancer is extremely poor. Although chemotherapy combined with immunotherapy has achieved promising efficacy in the first-line treatment of advanced gastric cancer, patients with peritoneal metastasis benefit less from this regimen. Hyperthermic intraperitoneal chemotherapy (HIPEC) represents a novel treatment option, which maintains the high concentration of drugs in the abdominal cavity, and improve the anti-tumor efficacy of chemotherapy drugs through the thermo-thermal effect. The purpose of this study is to investigate the efficacy and safety of HIPEC and systemic chemotherapy combined with sintilimab in the first-line treatment of advanced gastric cancer and gastroesophageal junction adenocarcinoma with peritoneal metastasis.

DETAILED DESCRIPTION:
To determine the efficacy and safety of HIPEC and systemic chemotherapy combined with sintilimab in the first-line treatment of advanced gastric cancer with peritoneal metastasis, patients will receive SOX regimen chemotherapy combined with sintilimab, once every three weeks. In the first cycle, HIPEC will be administrated, and HIPEC or intraperitoneal chemotherapy will be administrated in the second to third cycles according to the patient's condition. Then, another 3-cycle SOX regimen of systemic chemotherapy will be administrated. After the end of 6 cycles, patients will receive maintain treatment with a combination of S-1 and sintilimab until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Unresectable gastric/gastroesophageal junction adenocarcinoma diagnosed with peritoneal metastasis through laparoscopic exploration and pathological or cytological examination;
3. No previous antitumor treatment.
4. Agree to provide blood/tissue specimens.
5. The expected survival is more than 3 months.
6. ECOG PS≤1.
7. Adequate organ function including the following:

   1. Total bilirubin ≤1.5 times the upper limit of normal (ULN);
   2. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3×ULN;
   3. Alkaline phosphatase≤2.5×ULN (if the tumor invaded the liver, ≤3×ULN);
   4. Serum creatinine≤1.5×ULN;
   5. Serum amylase and lipase≤1.5×ULN;
   6. International standardized ratio (INR)/partial thromboplastin time (PTT)≤1.5×ULN;
   7. Platelet count ≥ 75,000 /mm3;
   8. Hemoglobin (Hb) ≥ 9 g/dL;
   9. Absolute neutrophil count (ANC) ≥ 1500/mm3;
8. Strict contraception.
9. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Undergoing other drug clinical trials or having participated in any drug clinical trials one month before enrollment.
2. Active autoimmune disease or history of refractory autoimmune disease.
3. Receiving corticosteroids (> 10mg/d prednisone or equivalent dose of steroids) or other systematic immunosuppression therapies within 14 days before enrollment, excluding the following therapies: steroid hormone replacement therapy (≤10mg/d); local steroid therapy; and short-term, prophylactic steroid therapy for preventing allergies or nausea and vomiting.
4. Active or clinically significant cardiac disease:

   1. Congestive heart failure > New York Heart Association (NYHA) class 2;
   2. Active coronary artery disease;
   3. Arrhythmias requiring treatment other than β-blockers or digoxin;
   4. Unstable angina (with angina symptoms at rest), new angina within 3 months before enrollment, or new myocardial infarction within 6 months before enrollment
5. Gastrointestinal perforation, obstruction, or uncontrollable diarrhea in the 6 months prior to enrollment;
6. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor was cured and no evidence of disease was found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
7. Patients with pheochromocytoma.
8. Patients with a history of HIV infection or active hepatitis B/C.
9. Ongoing > level 2 infection.
10. Symptomatic brain metastasis or meningioma.
11. Unhealed wounds, ulcers or fractures.
12. Renal failure patients requiring blood or peritoneal dialysis.
13. Epileptic that needs medication.
14. History of organ transplantation (including corneal transplantation).
15. Allergic to research drugs or similar drugs, or suspected allergies.
16. Pregnant or lactating women.
17. Medical, psychological or social conditions can affect the recruitment of patients and evaluation of study results.
18. Other antitumor therapy (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) other than investigator drugs. Palliative external irradiation for non-target lesions is allowed.
19. Previously used similar chemotherapy drugs or immune checkpoint inhibitors;
20. Major surgery 4 weeks before recruitment, open biopsy or major trauma surgery (excluding biliary stents, or percutaneous biliary drainage).
21. Treatment with antitumor Chinese herbal medicine.
22. Vaccination history 4 weeks prior to enrollment
23. The investigator believes that patients who are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every 3 month postoperation up to 24 months
  Overall survival (OS) is defined as the time from randomization to death

SECONDARY OUTCOMES:
ORR | every 3 month postoperation up to 24 months
  Objective Response Rate
DCR | every 3 month postoperation up to 24 months
  disease control rate
Progression-free survival | every 3 month postoperation up to 24 months
  Progression-free survival (PFS) is defined as the time from randomization to diesea progression
Safety and Tolerability | every 3 month postoperation up to 24 months
  Treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yang, M.D., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No